CLINICAL TRIAL: NCT01798368
Title: An Open Label Study to Evaluate the Safety and Tolerability of Nasal Stimulation Using the PBASE System in Non-patient Volunteers
Brief Title: PBASE-system Safety and Tolerability Clinical Investigation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PS002
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Non-patient Volunteers

ARMS (1):
- PBASE system 2.0 (Experimental)
  Interventions: Device: PBASE system 2.0

INTERVENTIONS:
Device: PBASE system 2.0

SUMMARY:
The purpose of this study is to demonstrate that the treatment does not cause any clinically significant effects that would put patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to participation in the clinical investigation
* Judged by the Investigator as suitable for participation in the study without safety concerns based on medical history, physical examination and laboratory results
* Age: 18-65 years of age.
* Gender: Male or female subjects.
* Negative urine drug screen (amphetamine, benzodiazepines, cocaine, marijuana, metamphetamine, morphine) at screening and Visit 2.
* Female subjects have to be post-menopausal for more than one year or use a highly efficient method of contraception (i.e. a method with less than 1% failure rate [e.g. sterilisation, hormone implants, hormone injections, some intrauterine devices, abstinence, or vasectomised partner]). Oral contraceptives: combined pill (estrogen / progestin) and medium-dose progestin pill (for example desogestrel 75ug) are accepted only in combination with the partner using condoms.
* Willing and able to comply with all study procedures and restrictions

Exclusion Criteria:

* A diagnosis of asthma or chronic obstructive pulmonary disorder.
* Ongoing respiratory infection including the nasal cavity.
* Current malignancy of any kind.
* History of frequent nose bleeds or a condition that increases the risk of excessive bleeding.
* Pronounced anterior septal deviation or other significant nasal pathology.
* Known allergy to polyvinylchloride or medicinal liquid paraffin.
* Ongoing treatment with drugs indicated for respiratory or cardiac disorders.
* Any disease, condition (medical or surgical) including allergic, immunological and gastro-intestinal conditions and/or chronic medications which, in the opinion of the investigator, might compromise the study results, or would place the subject at increased risk.
* Vital signs with clinically significant deviations that would make the subject unsuitable for the study, as judged by the investigator.
* Evidence of significant cardiovascular disease defined by the following:

  1. New York Heart Association (NYHA) Class III or IV heart failure;
  2. Presence of symptomatic coronary artery disease or unstable angina;
  3. Persistent arrhythmia requiring chronic pharmacotherapy or implantable device;
  4. Clinically significant abnormalities seen on the screening electrocardiogram as assessed by the investigator;
* Clinically significant deviations in, hematology (including coagulation parameters aPTT and INR) variables, blood chemistry variables or urinalysis as assessed by the investigator.
* Positive screening test for HIV or hepatitis B or C
* Positive alcohol breath test at Visit 1 or at Visit 2.
* Non-smoker since at least six months at time of screening.
* Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Previously treated with radiation on the face
* Previous radiation therapy to the head or neck regions
* Previously treated with an implantable stimulator or any implantable device in the head and / or neck
* Has a recent or repeated history of syncope.
* Has a recent or repeated history of seizures.
* Surgery within the past three months, determined by the PI to be clinically relevant.
* Strenuous exercise within 2 days of Visit 1 or Visit 2.
* Women who are pregnant or nursing.
* Female subjects: unwilling to use adequate contraceptive measures from the signing of the informed consent until end of the study at the follow-up visit.
* Received study drug in a clinical trial for an investigational drug within the previous 30 days, or 5 half-lives, whichever is longer.
* Blood donation or loss of whole blood exceeding 100 mL within 30 days from screening or plasma within 14 days from screening.
* Excessive intake of alcohol, defined as an average daily intake of greater than three units, or a maximum weekly intake of greater than 21 units ((three units equal 250 ml of 12% alcohol by unit wine).
* Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in ECG variables | Approximately 1 hour prior to treatment initiation to 3 hours post treatment termination
  ECG variables as documented on continuous recording include heart rate, heart rate variability,T-wave morphology, and occurrence of arrhythmias
Change in Vital signs | Approximately 1 hour prior to treatment initiation, right before treatment initiation, 10 min after treatment termination and 3 hours after treatment termination
  Vital signs measurements include blood pressure, pulse and respiratory rate